CLINICAL TRIAL: NCT01491854
Title: Long-term Safety Follow-up After Growth Hormone Treatment (rhGH) of Short Children Born Small for Gestational Age (SGA)
Brief Title: Long-term Safety Follow-up After Growth Hormone Treatment of Short Children Born Small for Gestational Age
Acronym: SGA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: in accordance with the request to close study EP00-402 "EMEA/H/C/000607/MEA 10.2" submitted and adopted by the EMA
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CEP00-402
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Short Children Born Small for Gestational Age (SGA)
Keywords: Long-term; safety; follow-up; growth hormone treatment; short children; Small for Gestational Age; Somatropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitoring of long-term safety (Other): Long-term safety follow-up after the end of treatment with Omnitrope (single arm)
  Interventions: Other: Bloodsampling

INTERVENTIONS:
Other: Bloodsampling — Bloodsampling

SUMMARY:
This study is performed as part of the Marketing Authorisation Holder's post-marketing pharmacovigilance plan to investigate the long-term safety, in particular the diabetogenic potential and immunogenicity of rhGH therapy in short children born small for gestational age (SGA).

DETAILED DESCRIPTION:
The purpose of this study is

1. to monitor short children born SGA who were treated with growth hormone in study EP00-401 for the development of diabetes for a further 10 years after termination of growth hormone treatment

   and
2. to report the incidence of anti-rhGH antibodies and of E. coli host cell peptide (HCP) antibodies (ABs) for 6 months after termination of GH treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients who fulfilled the diagnosis SGA, participated in study EP00-401, and received at least one dose of study medication
* Written informed consent of patient (for children who can read and/ or understand) and/or parent or legal guardian

Exclusion Criteria:

* Patients unwilling and/or parents/guardians who are not capable of ensuring compliance with the provisions of the study protocol

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-07-20 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz Biopharmaceuticals Sandoz, Study Chair — Sandoz GmbH
Locations (22):
- Czechia (3):
  - Novartis Investigative Site, Ústí nad Labem, Czech Republic
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Tbilisi, Georgia
- Germany (2):
  - Novartis Investigative Site, Nordrhein Westfalen, Sankt Augustin
  - Novartis Investigative Site, München
- Novartis Investigative Site, Miskolc, Hungary
- Poland (12):
  - Novartis Investigative Site, Poznai, Greater Poland Voivodeship
  - Novartis Investigative Site, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Novartis Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Novartis Investigative Site, Rzeszów, Podkarpackie Voivodeship
  - Novartis Investigative Site, Katowice, Silesian Voivodeship
  - Novartis Investigative Site, Zabrze, Silesian Voivodeship
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Kielce, Świętokrzyskie Voivodeship
- Romania (3):
  - Novartis Investigative Site, Lasi, Iaşi
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 130 participants signed informed consent. Of the 130 enrolled subjects, 11 subjects had no post-baseline visit, leading to exclusion from the SAF/FAS. Another subject was excluded as he received treatment with Omnitrope, which was not consistent with the protocol. Accordingly, 118 subjects comprised the SAF and in the FAS
Pre-assignment Details: SAF : safety Analysis set FAS : full Analysis set
Period: Overall Study
Arm/Group | Monitoring of Long-term Safety
Started | 130
Completed | 0
Not Completed | 130
Not completed — mainly due to premature termination | 93
Not completed — Death | 1
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 33

BASELINE CHARACTERISTICS:
Arm/Group | Monitoring of Long-term Safety
Number analyzed (Participants) | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.79 (2.848)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: full Analysis set
  Participants
    Female | 64
    Male | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Caucasian | 118

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Long-term Effect of Growth Hormone Treatment on the Development of Diabetes After End of Therapy.
Description: Number of participants diagnosed with Diabetes mellitus type 2 during the study, defined as fullfilment of these 3 criteria:
  * FPG ≥ 126 mg/dl (7.0 mmol/L) during blood sampling and/or during Oral Glucose Tolerance Test (OGTT)
  * 2-h plasma glucose ≥ 200 mg/dl (11.1 mmol/L) during an OGTT
  * Investigator documenting diagnosis of diabetes mellitus type 2 during OGTT
Time Frame: 5 years
Population: full Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Monitoring of Long-term Safety
Number analyzed (Participants) | 118
Participants | 0

2. Secondary Outcome: to Evaluate IGF-I and IGFBP-3 Levels After End of Growth Hormone Treatment
Time Frame: baseline, 6 months, 1 year , 5 years
Population: full Analysis set, with measure
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Monitoring of Long-term Safety
Number analyzed (Participants) | 118
nmol/L
  IGF-1 baseline: number analyzed (Participants) | 108
  IGF-1 baseline | 67.42 (31.137)
  IGF-1 6 months: number analyzed (Participants) | 95
  IGF-1 6 months | 48.42 (20.002)
  IGF-1 1 year: number analyzed (Participants) | 80
  IGF-1 1 year | 46.28 (21.555)
  IGF-1 5 years: number analyzed (Participants) | 12
  IGF-1 5 years | 44.60 (16.035)
  IGFBP-3 baseline: number analyzed (Participants) | 110
  IGFBP-3 baseline | 211.12 (49.523)
  IGFBP-3 6 months: number analyzed (Participants) | 95
  IGFBP-3 6 months | 187.79 (42.999)
  IGFBP-3 1 year: number analyzed (Participants) | 82
  IGFBP-3 1 year | 186.59 (47.246)
  IGFBP-3 5 years: number analyzed (Participants) | 13
  IGFBP-3 5 years | 180.00 (26.470)

3. Secondary Outcome: To Evaluate the Incidence of Anti-rhGH Antibodies After Termination of Growth Hormone Treatment.
Description: number of participants with positive results for anti-drug antibody (ADA). Percentages indicated are calculated based on the total number of patients (118 participants).
Time Frame: baseline, 6 months, 1 year, 5 years
Population: safety Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Monitoring of Long-term Safety
Number analyzed (Participants) | 118
Participants
  baseline: number analyzed (Participants) | 110
  baseline | 0
  6 months: number analyzed (Participants) | 91
  6 months | 1
  1 year: number analyzed (Participants) | 2
  1 year | 0
  5 years: number analyzed (Participants) | 0
  5 years | 0

4. Primary Outcome: To Evaluate the Long Term Effects of rhGH on Carbohydrate Metabolism Through Fasting Plasma Glucose (FPG) Levels
Description: Supportive to Primary Endpoint
Time Frame: baseline, 6 months, 1 year, 5 years
Population: safety Analysis set with measure
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Monitoring of Long-term Safety
Number analyzed (Participants) | 118
mmol/L
  FPG baseline: number analyzed (Participants) | 109
  FPG baseline | 4.69 (0.492)
  FPG 6 months: number analyzed (Participants) | 90
  FPG 6 months | -0.13 (0.567)
  FPG 1 year: number analyzed (Participants) | 79
  FPG 1 year | -0.14 (0.457)
  FPG 5 years: number analyzed (Participants) | 11
  FPG 5 years | -0.37 (0.856)

5. Primary Outcome: To Evaluate the Long Term Effects of rhGH on Carbohydrate Metabolism Through Fasting Insulin Levels
Description: Supportive to Primary Endpoint
Time Frame: baseline, 6 months, 1 year, 5 years
Population: full Analysis set with measure
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Monitoring of Long-term Safety
Number analyzed (Participants) | 118
pmol/L
  baseline: number analyzed (Participants) | 109
  baseline | 70.87 (38.477)
  6 months: number analyzed (Participants) | 88
  6 months | -2.34 (38.267)
  1 year: number analyzed (Participants) | 75
  1 year | -7.48 (34.676)
  5 years: number analyzed (Participants) | 12
  5 years | 3.40 (52.526)

6. Primary Outcome: To Evaluate the Long Term Effects of rhGH on Carbohydrate Metabolism Through Glucose Glycolsylated Hemoglobin (HbA1c)
Description: Supportive to Primary Endpoint
Time Frame: baseline, 6 months, 1 year, 5 years
Population: full Analysis set with measure
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Monitoring of Long-term Safety
Number analyzed (Participants) | 118
percentage
  baseline: number analyzed (Participants) | 107
  baseline | 5.280 (0.3569)
  6 months: number analyzed (Participants) | 87
  6 months | -0.057 (0.3621)
  1 year: number analyzed (Participants) | 78
  1 year | -0.108 (0.2931)
  5 years: number analyzed (Participants) | 12
  5 years | -0.308 (0.6036)

7. Secondary Outcome: to Evaluate Final Height
Time Frame: baseline, 6 months, 1 year, 5 years
Population: Full Analysis set with measure
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Monitoring of Long-term Safety
Number analyzed (Participants) | 118
cm
  baseline: number analyzed (Participants) | 115
  baseline | 152.63 (16.362)
  6 months: number analyzed (Participants) | 99
  6 months | 152.41 (16.894)
  1 year: number analyzed (Participants) | 88
  1 year | 152.43 (16.698)
  5 years: number analyzed (Participants) | 13
  5 years | 150.42 (12.938)

8. Primary Outcome: To Evaluate the Long Term Effects of rhGH on Carbohydrate Metabolism Through HOMA and QUICKI Scores
Description: Supportive to Primary Endpoint. HOMA = homeostasis model assessment for Insulin resistance: Healthy Range: 1.0 (0.5-1.4).
  < 1.0 means you are insulin-sensitive which is optimal. >1.9 indicates early insulin resistance. > 2.9 indicates significant insulin resistance. The quantitative insulin sensitivity check index (QUICKI) measures insulin sensitivity, which is the inverse of insulin resistance. The QUICKI calculation for insulin resistance in humans fall broadly within a range between 0.45 for unusually healthy individuals and 0.30 in diabetics. Lower numbers reflect greater insulin resistance.
Time Frame: baseline, 6 months, 1 year, 5 years
Population: safety Analysis set with measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monitoring of Long-term Safety
Number analyzed (Participants) | 118
score on a scale
  HOMA score baseline: number analyzed (Participants) | 107
  HOMA score baseline | 2.082 (1.0336)
  HOMA score 6 months: number analyzed (Participants) | 86
  HOMA score 6 months | -0.073 (1.1447)
  HOMA score 1 year: number analyzed (Participants) | 73
  HOMA score 1 year | -0.206 (1.0170)
  HOMA score 5 years: number analyzed (Participants) | 11
  HOMA score 5 years | 0.094 (1.8835)
  QUICKI score baseline: number analyzed (Participants) | 107
  QUICKI score baseline | 0.354 (0.0459)
  QUICKI score 6 months: number analyzed (Participants) | 86
  QUICKI score 6 months | 0.004 (0.0350)
  QUICKI score 1 year: number analyzed (Participants) | 73
  QUICKI score 1 year | 0.012 (0.0413)
  QUICKI score 5 years: number analyzed (Participants) | 11
  QUICKI score 5 years | 0.022 (0.0703)

ADVERSE EVENTS:
Time Frame: approximately 9 years
Description: AE additional description
Groups:
- Total: Total
Arm/Group | Total
All-Cause Mortality (participants affected / at risk) | 1/118
Serious Adverse Events (participants affected / at risk) | 8/118
Other Adverse Events (participants affected / at risk) | 23/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=118)
Anaemia (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Chronic tonsillitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Epilepsy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
VIth nerve paralysis (Nervous system disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Oligomenorrhoea (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total (N=118)
Hypothyroidism (Endocrine disorders) | 4
Nasopharyngitis (Infections and infestations) | 7
Pharyngitis (Infections and infestations) | 5
Respiratory tract infection (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Headache (Nervous system disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 4

LIMITATIONS AND CAVEATS:
The study was terminated prematurely in accordance with the request to close study EP00-402 "EMEA/H/C/000607/MEA 10.2" submitted to the EMA on 29-Mar-2018 and adopted by the EMA on 28-Jun-2018

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2014-07-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT01491854/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT01491854/SAP_001.pdf